CLINICAL TRIAL: NCT05747833
Title: Randomized Controlled Trial: The Effect of Preparation for Procedure With Toy IV Catheter Before Peripheral Cannula Administration on Children's Pain, Fear, and Emotional Indicators
Brief Title: The Effect of Toy IV Catheter on Children's Pain, Fear and Emotional Indicators
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, Hazal USLU, Nurse, Eskisehir Osmangazi University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 10346826
Record Dates: First submitted 2022-12-26; First posted 2023-02-28 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Intravenous Catheterization
Keywords: Toy; Therapeutic play; Preparation; Pain; Fear
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Toy IV Catheter Before Peripheral Cannula application (Experimental): Intervention Group: Child Fear Scale will be applied to the children who will meet the inclusion criteria. The data collection form will be filled in by the researcher according to the information received from the patient file and parents. Children in the intervention group will be shown the procedure on the doll with the IV Catheter developed by the researchers, and then it will be applied to it.
  Interventions: Other: Children Preparation With a Toy IV Catheter Before Peripheral Cannula application
- Standard of care (No Intervention): Control group will not be aplied other than the normal procedure of the hospital. In both groups, at the end of the procedure, the child's reactions will be observed during the procedure and the Wong-Baker Faces Pain Scale, the Child Anxiety Scale and the Child Emotional Indicators Scale will be filled independently by the researcher and the parent in line with the child's reactions.

INTERVENTIONS:
Other: Children Preparation With a Toy IV Catheter Before Peripheral Cannula application — THE EFFECT OF PROCESSING PREPARATION WITH A TOY IV CATHETER BEFORE PERIPHERAL CANNULA APPLICATION ON CHILDREN'S PAIN, FEAR and EMOTIONAL INDICATORS
  Arms: Toy IV Catheter Before Peripheral Cannula application

SUMMARY:
Aim: Research was conducted to determine the effect of preparation for the procedure with a toy IV catheter before IV catheterization in children aged 6-10 years, on children's pain, fear and emotional indicators.

Methods: It is a randomized controlled intervention study. The study was completed with 80 children. There are two groups in the study. Before the IV catheterization, the children in the intervention group were treated with the toy IV catheter developed by the researchers on the knitted doll, and then the procedure was provided to them. Conversely, no intervention was applied to the control group other than the normal procedure of the hospital. Stratified block randomization method was used to assign children to groups. In the study; "Personal Data Collection Form", "Wong-Baker Faces Pain Scale (WBFPS)", "Child Fear Scale (CFS)" and "Child Emotional Manifestation Scale (CEMS)" were used to collect data.

DETAILED DESCRIPTION:
Children may be sick during their normal development and may have to come to the hospital. For children, the hospital environment, especially emergency rooms, conveys uncertainty. The reason for this uncertainty; the presence of health team members that children do not know, equipment they have not seen before, and interventions. The child's sense of uncertainty and the thought that his own control is in danger may cause him to become stressed and afraid of the hospital. As a matter of fact, studies on children's hospital experience indicate that they experience negative emotions such as stress, anger, restlessness, and tension. It is known that the most common negative emotion and experience children experience in the hospital environment is anxiety due to pain and fear.

Children can experience pain in all healthcare settings. Almost all diagnostic and therapeutic applications cause pain. It is also known that children experience more fear in the hospital environment than adults. Among the biggest fears children experience in the hospital environment are; Losing body functions, having surgery can be counted as painful invasive procedures performed for diagnosis and treatment. Especially made using a needle such as an injector; Procedures such as vaccination, bloodletting, and IV catheterization may cause pain and fear in children.

More than 80% of children admitted to hospitals are administered IV catheters. Almost all children are adversely affected by this process. In reducing these negative emotions experienced, it is very important to prepare children for the procedure. Control of pain and fear; requires cooperation between physicians, nurses and other health professionals. Especially nurses have important duties in this regard, as they have the opportunity to observe the patient closely and for a longer period of time. The American Association of Pain Management Nursing (ASPMN) also reports that nurses are responsible for controlling pain using pharmacological and non-pharmacological methods before, during and after painful intervention. For this purpose, therapeutic play can be used.

Therapeutic play is a type of play used to reduce the child's fear and stress towards the hospital, to alleviate the feeling of uncertainty, to evaluate misunderstandings about the hospital environment and the interventions applied in the hospital, to teach clinical procedures and to reduce pain in painful procedures. Ensuring that the child touches the tools and equipment to be used in the treatment during the game played in the hospital allows him to recognize them and perceive them as less threatening. At the same time, it improves the feeling of trust towards the health professional. Particularly, when preparation for play-based treatment is combined with treatment, the child can better tolerate painful procedures by developing positive coping methods. As a matter of fact, in the experimental study of Uluışık (2019) with 60 children aged 5-6 years, it was seen that the information provided with the play dough consisting of a dentist set reduced dental fear. In a randomized controlled study conducted by Miller et al. (2016) with 98 children aged 3-12, using an electronic device called Ditto (Diversionary Therapy Technologies, Brisbane, Australia) that provides procedural preparation and distraction during the vascular access procedure, significantly reduced stress. In another study conducted by Tunç Tuna and Açikgoz (2015) on 60 children aged 9-12, it was found that pre-procedural information on preparation for the peripheral venous cannula application in children and performing the procedure by showing it on the toy reduced the child's pain and anxiety. In the study conducted by Tunç Tuna and Açikgöz, real IV catheters were used in preparation for the procedure before the peripheral cannula application of the children. However, giving such tools and equipment to the hands of especially small children and having them applied can be dangerous and harmful for them. Instead, alternative methods should be developed.For example, the process can be explained through pictures and/or the toys/models of the tools to be used in the process can be given to children and practice can be made. In the literature review, no study could be found on the preparation of the child for the procedure with realistic toys before the IV catheterization procedure.

ELIGIBILITY:
Inclusion Criteria:

* Your child;
* Age between 6-10,
* To receive IV treatment upon the request of a physician,
* Being conscious and able to communicate verbally,
* Understanding and speaking Turkish,
* Having a mother and / or father with him,
* After the information, the child and his parents agree to participate in the study in writing and verbally,
* Pediatric Emergency Clinic has been accepted to the Green Area,
* Not using analgesic and / or sedative drugs in the last 8 hours.

Exclusion Criteria:

* Your child;
* Being younger than 6 and over 10 years old,
* Having pain,
* Having a high fever (body temperature of 38 ° C and above) Applying to the hospital with a complaint that requires urgent intervention such as convulsion or trauma,
* Having applied to the hospital by ambulance,
* Admitted to the Yellow or Red Area of the Pediatric Emergency Clinic after triage,
* Having had an IV catheter before,
* Having mental disability,
* Having a chronic and / or fatal disease, Having a diagnosis made by psychiatry,
* Communication problems with his family and / or himself (not speaking Turkish, agitation, etc.)

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2020-07-14 (Actual); Primary Completion 2022-05-15 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Personal data collection form | 1.5 month
  The data collection form was prepared by the researchers in line with the literature (Başkaya, 2019; Gültekin, 2019; Szeszak et al., 2016; Tunç Tuna & Açıkgoz 2015). In this form, 3 including the personal characteristics of the child, 9 questioning the illness and hospital experiences; There are 22 questions in total, 10 of which include parent and family characteristics.
Wong-Baker faces pain scale | 1.5 month
  The scale is based on measuring the level of pain by scoring facial expressions of children aged 3-18. There is a numerical value for each facial expression in the scale. This numerical value gives us information about the child's pain level. The lowest numerical value is "0" and the highest numerical value is "5". A high score on the scale indicates a high level of pain. The application of the scale is quite simple. Faces and numbers are explained to the child and asked to choose the face that best expresses his or her pain. This scale was used by the researcher to evaluate the pain of children before the procedure. In addition, in order to determine the pain felt by the child during the procedure after the procedure, it was filled out independently by the child, parent and researcher.
Child Fear Scale | 1.5 month
  The scale was developed by Mc Murtry et al. in 2011 to determine the anxiety level of children aged 5-10 years. There are various facial expressions in the scale and a numerical value is given for each facial expression. The lowest score obtained from the scale is "0" and the highest score is "4". The higher the score obtained from the scale, the higher the level of anxiety felt in the child. This scale was used by the researcher, parent and child to evaluate the anxiety of children before the procedure. After the procedure, it was filled again independently by the child, parent and researcher to determine the anxiety felt by the child during the procedure.
Child Emotional Manifestation Scale | 1.5 month
  In the scale, emotional indicators are evaluated in terms of 5 parameters. These parameters are; facial expression, voice, activity, interaction and cooperation level. These five parameters are scored from 1 to 5, and the lowest "5" and the highest "25" points are obtained at the end of the evaluation of the scale. A low score from the scale indicates a positive emotional state, and an increase in a score indicates a negative emotional state. This scale was filled in independently by the parent and the researcher in order to evaluate the emotional indicators of the child during the procedure after the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Hazal USLU, Study Director — Eskişehir Osmangazi University
Locations (1):
- Hazal, Eskişehir, Odunpazarı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No